CLINICAL TRIAL: NCT05538741
Title: Comparison of the Incidence of Hypotension with Bolus Versus Continuous Remimazolam for Anesthetic Induction in Elderly Patients
Brief Title: Hypotension After Anesthetic Induction with Remimazolam in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RMZ_bolcon_old
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bolus (Experimental): Remimazolam bolus injection for 20 seconds
  Interventions: Drug: Bolus of remimazolam
- Continuous (Active Comparator): Remimazolam continuous infusion
  Interventions: Drug: Continuous infusion of remimazolam

INTERVENTIONS:
Drug: Bolus of remimazolam — 0.19-0.25 mg/kg for 60-80 years old 0.14-0.19 mg/kg for >80 years old
  Arms: Bolus
Drug: Continuous infusion of remimazolam — 12 mg/kg/hr until loss of consciousness
  Arms: Continuous

SUMMARY:
Even though remimazolam is known to be safely administered without hemodynamic instability, hypotension is the one of the common side effects of remimazolam. Because elderly patients are susceptible to hypotension due to old age, multimodality, and multiple medications, hypotension can be harmful in elderly patients. Remimazolam can be administered either bolus or continuous for anesthetic induction. In our study the investigators aimed to compare the incidence of hypotension after anesthetic induction using remimazolam by bolus injection and continuous infusion in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with age over 60 years old
* scheduled for elective surgery under general anesthesia
* American Society of Anesthesiology Physical Status I-III

Exclusion Criteria:

* Arrhythmia
* Liver dysfunction
* Kidney dysfunction
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Allergic to benzodiazepines
* Heart failure
* Drug intoxication
* Alcoholics
* Cognitive dysfunction
* Unable to understand and consent voluntarily

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
The incidence of hypotension | 10 minutes after intubation
  Systolic blood pressure < 90 mmHg

SECONDARY OUTCOMES:
The incidence of bradycardia | 10 minutes after intubation
  Heart rate < 40 beats per minute
Number of participants with use of any vasopressors | 10 minutes after intubation
  Use of ephedrine, phenylephrine
Lowest systolic blood pressure | 10 minutes after intubation
  The lowest systolic blood pressure measured within10 minutes after intubation
Time to loss of consciousness | 10 minutes after intubation
  Time to loss of consciousness. Loss of consciousness is assessed by the loss of response to shoulder shaking.
Total remimazolam used for anesthetic induction | 10 minutes after intubation
  Sum of remimazolam used during anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided